CLINICAL TRIAL: NCT05876169
Title: How Does Orthognathic Surgery Affect Jaw and Neck Motor Function?
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-kakfunktion
Record Dates: First submitted 2023-05-02; First posted 2023-05-25 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Cleft Lip and Palate
Keywords: Orthognathic Surgery; Cleft Lip and Palate
MeSH Terms: conditions — Cleft Lip | interventions — Orthognathic Surgery; Head Movements; Bite Force

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prospective longitudinal study design (Other): Patients that will undergo orthognatic surgery will be given opportunity to participate in jaw and neck motor function analysis.
  Interventions: Procedure: Orthognathic surgery

INTERVENTIONS:
Procedure: Orthognathic surgery — Surgical corrections of the maxilla and/or the mandible. Integrated jaw-neck movement patterns, muscle activity, bite force and occlusal contact area will be registered and mapped with quantitative objective functional variables. The state-of-the-art core equipment to evaluate jaw-neck motor function in detail is located in the Movement Lab (Department of Odontology, Umeå University).
  Other Names: Kinematic of jaw and head movements, muscle activity, bite force, occlusal contact area

SUMMARY:
In a prospective longitudinal study design, details in jaw-neck kinematics and electromyography (EMG) activity changes in patients (women and men) referred for surgical correction of basal relations between the maxilla and mandible over time; pre-operative and during follow-up 8 weeks and 18 months after surgical correction will be evaluated. The results will contribute with novel insights on jaw-neck motor function before, in short- and long-term after the surgical process. We will have blinded evaluation of outcomes.

DETAILED DESCRIPTION:
Consecutive patients referred to department of Oral and Maxillofacial Surgery, Umeå University Hospital for corrective maxillofacial-mandibular surgery, will offer opportunity to be included in the study. Expected number of patients: 20 - 25 patients annually. Blinded evaluation will be pre-operative and during follow-up 8 weeks and 18 months after surgical correction.

ELIGIBILITY:
Inclusion Criterias:

* Patients accepted for orthognathic surgery due to jaw discrepancies.
* Patients given their consent for participation

Exclusion Criterias:

* Patients with syndromes
* Patients not given their consent for participation
* Patients unable to follow instructions due to lack of knowledge in Swedish and/or English language

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-09-06 (Actual); Primary Completion 2026-12-12 (Estimated); Study Completion 2026-12-12 (Estimated)

PRIMARY OUTCOMES:
Change in Kinematic outcome variables | Preoperatively, postoperatively 8 weeks, 18 months
  Jaw and head movement amplitudes (mm)
Change in Kinematic outcome variables | Preoperatively, postoperatively 8 weeks, 18 months
  Movement cycle time (s)
Change in Kinematic outcome variables | Preoperatively, postoperatively 8 weeks, 18 months
  Movement acceleration from start to peak (mm/s2)
Change in Kinematic outcome variables | Preoperatively, postoperatively 8 weeks, 18 months
  Jaw movement area (mm2)
Change in Kinematic outcome variables | Preoperatively, postoperatively 8 weeks, 18 months
  Jaw movement volume (mm3)
Change in Electromyography (EMG) | Preoperatively, postoperatively 8 weeks, 18 months
  Muscle activity in micro-Volt in jaw and neck muscles bilaterally
Change in Maximum voluntary occlusal bite force (MVOBF) | Preoperatively, postoperatively 8 weeks, 18 months
  Newton (N)
Change in Occlusal contact area | Preoperatively, postoperatively 8 weeks, 18 months
  mm2

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Department of Odontology, Umeå University, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: No